CLINICAL TRIAL: NCT04881682
Title: Immunoadsorption Versus Immunoglobulins for Treatment of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Acronym: IVITOC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IVITOC 1.1
Record Dates: First submitted 2021-04-28; First posted 2021-05-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: CIDP
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Plasmapheresis; Immunoglobulins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunoadsorption (Experimental): 3 cycles of immunoadsorption in week 1, 7, and 13 after randomization. One cycle consists of 5 sessions on 5 consecutive days with processing of the 2-fold plasma volume on the first day and the 2.5-fold plasma volume on consecutive days, using regenerative adsorbers (Therasorb, Miltenyi Biotec, Bergisch Gladbach)
  Interventions: Device: Immunoadsorption
- Immunoglobulins (Active Comparator): 5 cycles of intravenous immunoglobulins in week 1, 4, 7, 10, and 13 after randomization. The first cycle consists of 5 intravenous applications of immunoglobulins on 5 consecutive days in a dosage of 0.4 g per kg body weight per day. Subsequent cycles consist of 2 intravenous applications of immunoglobulins on 2 consecutive days in a dosage of 0.5 g per kg body weight per day.
  Interventions: Biological: Immunoglobulins

INTERVENTIONS:
Device: Immunoadsorption — see arm/group description
  Arms: Immunoadsorption
Biological: Immunoglobulins — see arm/group description
  Arms: Immunoglobulins

SUMMARY:
This is a randomized controlled study evaluating safety and efficacy of repeated immunoadsorption versus immunoglobulins in steroid-refractory Chronic Inflammatory Demyelinating Polyneuropathy (CIDP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, probable, or definite CIDP (typical or atypical) according to European Federation of Neurological Societies (EFNS) guidelines
* Disease duration of 3 years or less
* Age 18 years or above
* Previous treatment with methyl-prednisolone and insufficient therapeutic response as judged by the treating physician, or contraindications against methyl-prednisolone, or clinically significant side effects under methyl-prednisolone therapy as judged by the treating physician

Exclusion Criteria:

* Clinical or laboratory evidence of manifest systemic infection, i.e., C-reactive protein (CRP) above 20 mg/l, or evidence of nitrite-positive urinary tract infection
* Intake of angiotensin converting enzyme inhibitor within 1 week before first treatment
* immunoglobulin A deficiency
* Other contraindications against immunoadsorption or intravenous immunoglobulins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
CIDP Score | 15 weeks
  The CIDP Score is a combined score of Inflammatory Cause and Treatment (INCAT) Disability Score, Oxford Muscle Strength Score, and Vibration Score, with each subscore equally weighted.
Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Score | 15 weeks
  Standard clinical score for CIDP, quantifying disability.
Oxford Muscle Strength Score (Medical Research Council, MRC) | 15 weeks
  Standard clinical score for evaluation of muscle strength / paresis. Muscle strength is evaluated on a scale between 0/5 (no movement) and 5/5 (full strength) at 8 pre-defined muscles (one proximal and one distal muscle at each extremity).
Vibration Score | 15 weeks
  Standard clinical score for evaluation of pallesthesia, using a 256 Hz tuning fork. The individual perception threshold for vibration sensations on a scale between 0/8 (no perception) and 8/8 (normal perception) will be determined at 4 predefined spots (processus styloideus radii and malleolus lateralis on each side).

SECONDARY OUTCOMES:
CIDP Score | 1, 7, and 13 weeks
  The CIDP Score is a combined score of Inflammatory Cause and Treatment (INCAT) Disability Score, Oxford Muscle Strength Score, and Vibration Score, with each subscore equally weighted.
Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Score | 1, 7, and 13 weeks
  Standard clinical score for CIDP, quantifying disability.
Oxford Muscle Strength Score (Medical Research Council, MRC) | 16 weeks
  Standard clinical score for evaluation of muscle strength / paresis. Muscle strength is evaluated on a scale between 0/5 (no movement) and 5/5 (full strength) at 8 pre-defined muscles (one proximal and one distal muscle at each extremity).
Vibration Score | 16 weeks
  Standard clinical score for evaluation of pallesthesia, using a 256 Hz tuning fork. The individual perception threshold for vibration sensations on a scale between 0/8 (no perception) and 8/8 (normal perception) will be determined at 4 predefined spots (processus styloideus radii and malleolus lateralis on each side).
Pain | 1, 7, 13, and 15 weeks
  Quantifying pain on a Visual Analog Scale between 0 (no pain) and 10 (maximum pain).
N20 Latency | 15 weeks
  N20 latency of Nervus medianus (both sides) in somatosensory evoked potentials (SEPs).
P40 Latency | 15 weeks
  P40 latency of Nervus tibialis (both sides) in somatosensory evoked potentials (SEPs).
Nerve Conduction Velocity | 15 weeks
  Nerve conduction velocities of clinically affected nerves as measured by electroneurography (ENG).
Euro Quality of Life 5 Dimension 5 Levels (EQ-5D-5L) | 1, 7, 13, and 15 weeks
  Quality of Life Scale
Immunoglobulin A | 1, 7, 13, and 15 weeks
  Immunoglobulin A serum levels
Immunoglobulin G | 1, 7, 13, and 15 weeks
  Immunoglobulin G serum levels
Immunoglobulin M | 1, 7, 13, and 15 weeks
  Immunoglobulin M serum levels
Interleukin-1 | 1, 7, 13, and 15 weeks
  Interleukin-1 serum levels
Interleukin-6 | 1, 7, 13, and 15 weeks
  Interleukin-6 serum levels
Anti-contactin-1 | 1, 7, 13, and 15 weeks
  Anti-contactin-1 serum levels
Anti-neurofascin155 | 1, 7, 13, and 15 weeks
  Anti-neurofascin155 serum levels
Anti-contactin-associated-protein1 | 1, 7, 13, and 15 weeks
  Anti-contactin-associated-protein1 serum levels
Anti-neurofascin186 | 1, 7, 13, and 15 weeks
  Anti-neurofascin186 serum levels
Anti-neurofascin140 | 1, 7, 13, and 15 weeks
  Anti-neurofascin140 serum levels
Neurofilament Light Chain (NfL) | 1, 7, 13, and 15 weeks
  Neurofilament light chain (NfL) serum levels
Therapeutic Response | 15 weeks
  Share of patients with at least 10% improvement in CIDP score compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Dorst, Prof, Principal Investigator — University of Ulm
Locations (1):
- Department of Neurology, University of Ulm, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, and figures), as well as the study protocol will be available. Data will be available beginning 3 months and ending 5 years following article publication. Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims in the approved proposal. Proposals should be directed to johannes.dorst@uni-ulm.de; to gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at https://www.uniklinik-ulm.de/neurologie.html.
Supporting Information: Study Protocol
Time Frame: 3 months after publication until 5 years after publication
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims in the approved proposal.
URL: https://www.uniklinik-ulm.de/neurologie.html